CLINICAL TRIAL: NCT01249521
Title: Open Label Phase II Study Evaluating the Combination of Bevacizumab and AMG386 Without Chemotherapy as First Line Treatment of Advanced Colorectal Cancer
Brief Title: Dual Targeting of Vascular Endothelial Growth Factor-A Together With Angiopoietins in Chemotherapy-naïve Metastatic Colorectal Cancer
Acronym: Vengeance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Austin Health (Other Government)
Responsible Party: Niall Tebbutt, Austin Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03501
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trebananib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AMG386 and bevacizumab — AMG386 10mg/kg qw iv Bevacizumab 7.5mg/kg q3w iv

SUMMARY:
This is a clinical trial investigating the effectiveness and safety of the combination of the study drugs bevacizumab and AMG386 in patients with advanced (metastatic) chemotherapy-naive bowel (colorectal) cancer. Chemotherapy has a significant impact in metastatic bowel cancer in terms of maintenance of quality of life and extension of survival. However, ultimately tumours will develop resistance to these agents and further treatment options are urgently required.

Angiogenesis is a process that results in the formation of new blood vessels. Similar to normal tissues, solid tumours require new blood vessels for growth and survival. Hence, drugs targeting angiogenesis may be useful treatment options for patients with bowel cancer.

AMG386 and bevacizumab act on 2 different pathways relevant to angiogenesis. There is evidence from laboratory and animal studies to suggest that such a combination could be useful as a cancer treatment. Previous studies in humans have shown that AMG386 and bevacizumab can be combined safely.. This study aims to evaluate the effectiveness and safety of the combination of AMG386 and bevacizumab in patients with advanced bowel cancer.

40 patients from approximately four hospitals in Australia will participate in this trial, with approximately 20 patients being enrolled at Austin Health. All participants will receive the same treatment.

ELIGIBILITY:
Inclusion Criteria:

i) Histological diagnosis of colorectal cancer ii) Metastatic disease that is not resectable iii) Age > 18 years iv) Any patient in whom the investigator considers immediate cytotoxic chemotherapy is not required.

v) Measurable and/or non-measurable disease as assessed by CT scan vi) ECOG performance status 0, 1 or 2. vii) No prior chemotherapy except for adjuvant chemotherapy. viii) Adequate bone marrow function with platelets > 100 X 109/l; neutrophils > 1.5 X 109/l ix) Adequate renal function, with calculated creatinine clearance >40 ml/min (Cockcroft and Gault).

x) Adequate hepatic function with serum total bilirubin < 1.5 X upper limit of normal range xi) Life expectancy of at least 12 weeks xii) No other concurrent uncontrolled medical conditions xiii) No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other cancer treated with curative intent >2 years previously without evidence of relapse xiv) Women and partners of women of childbearing potential must agree to use adequate contraception xv) Written informed consent including consent for biomarker studies

Exclusion Criteria:

i) Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol ii) Uncontrolled hypertension iii) Prior treatment with VEGF inhibitors or angiopoietin inhibitors iv) Active bleeding disorders within the last 6 months v) Participation in any investigational drug study within the previous 4 weeks vi) Patients with uncontrolled clinically significant cardiac disease, arrhythmias or angina pectoris vii) Patients with a history of arterial or venous thrombosis within the last 12 months viii) Concurrent or prior (within 1 week before enrollment) anticoagulation therapy. The concurrent use of low molecular weight heparin or low dose warfarin (ie, 1 mg daily) for prophylaxis against thrombosis is acceptable while on study ix) Regular use of aspirin (>325mg/day) or NSAIDs (low dose aspirin (<325 mg/d), or occasional use of NSAIDs is acceptable) x) Treatment with immune modulators such as cyclosporine or tacrolimus within the previous 4 weeks xi) CNS metastases xii) Major surgical procedure within the last 28 days xiii) Minor surgical procedure, placement of access device, or fine needle aspiration within the last 7 days xiv) Serious non-healing wound, ulcer or bone fracture xv) 24 hour urinary protein > 1g/ 24 hours ( performed if urine dipstick > 1+ ) xvi) Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Disease control (ie non progression) at 6 months | 6 months

SECONDARY OUTCOMES:
Toxicity | weekly
Overall survival | 3 monthly
Response rate | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Niall Tebbutt, Study Chair — Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia